CLINICAL TRIAL: NCT06627556
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Single and Multiple Ascending Doses of H021 in Healthy Participants
Brief Title: A Study of Single and Multiple Ascending Doses of H021 in Healthy Participants
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu Carephar Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KFP-2024-H021-HW-101
Record Dates: First submitted 2024-10-03; First posted 2024-10-04 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-09

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (10):
- SAD Cohort 1: H021 6.25 milligrams (mg) (Experimental): Participants will receive H021, 6.25 mg oral tablet, as single-dose on Day 1 under fasting or fed conditions.
  Interventions: Drug: H021
- SAD Cohort 2: H021 12.5 mg (Experimental): Participants will receive H021, 12.5 mg oral tablet, as single-dose on Day 1 under fasting conditions.
  Interventions: Drug: H021
- SAD Cohort 3: H021 25 mg (Experimental): Participants will receive H021, 25 mg oral tablet, as single-dose on Day 1 under fasting conditions.
  Interventions: Drug: H021
- SAD Cohort 4: H021 50 mg (Experimental): Participants will receive H021, 50 mg oral tablet, as single-dose on Day 1 under fasting conditions.
  Interventions: Drug: H021
- SAD Cohort 5: H021 100 mg (Experimental): Participants will receive H021, 100 mg oral tablet, as single-dose on Day 1 under fasting conditions.
  Interventions: Drug: H021
- MAD Cohort 6: H021 12.5 mg (Experimental): Participants will receive H021, 12.5 mg oral tablet once daily from Day 1 to Day 7 under fasting conditions.
  Interventions: Drug: H021
- MAD Cohort 7: H021 25 mg (Experimental): Participants will receive H021, 25 mg oral tablet once daily from Day 1 to Day 7 under fasting conditions.
  Interventions: Drug: H021
- MAD Cohort 8: H021 50 mg (Experimental): Participants will receive H021, 50 mg oral tablet once daily from Day 1 to Day 7 under fasting conditions.
  Interventions: Drug: H021
- SAD-H021 Placebo (Placebo Comparator): Participants will receive H021, placebo oral tablet, as single-dose on Day 1 under fasting or fed conditions.
  Interventions: Drug: H021 Placebo
- MAD-H021 Placebo (Placebo Comparator): Participants will receive H021, placebo oral tablet once daily from Day 1 to Day 7 under fasting conditions.
  Interventions: Drug: H021 Placebo

INTERVENTIONS:
Drug: H021 — H021 oral tablet.
  Arms: MAD Cohort 6: H021 12.5 mg; MAD Cohort 7: H021 25 mg; MAD Cohort 8: H021 50 mg; SAD Cohort 1: H021 6.25 milligrams (mg); SAD Cohort 2: H021 12.5 mg; SAD Cohort 3: H021 25 mg; SAD Cohort 4: H021 50 mg; SAD Cohort 5: H021 100 mg
Drug: H021 Placebo — H021 placebo oral tablet.
  Arms: MAD-H021 Placebo; SAD-H021 Placebo

SUMMARY:
The primary purpose of this study is to evaluate the safety and tolerability of H021 tablets following oral administration of single and multiple ascending doses in healthy participants.

DETAILED DESCRIPTION:
This is a single center, Phase 1, randomized, double-blind, placebo controlled, sequential single ascending dose/multiple ascending dose (SAD/MAD) study, with a food-effect arm. The study will be divided into two parts:

* SAD cohorts, with food-effect evaluation
* MAD cohorts The two parts will be completed sequentially but with partial overlapping. The MAD phase can start once safety, tolerability, and pharmacokinetic data from the SAD phase show that single doses of at least 25 mg are acceptable. If the 25 mg dose will be not reached in the SAD phase, the Safety Review Committee (SRC) will set a new starting dose.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, non-smoker (no use of tobacco or nicotine products within 3 months prior to screening), greater than and equal to (>=) 18 and less than and equal to (<=) 55 years of age, with body mass index (BMI) greater than (>)18.5 and less than (<) 32.0 kilograms per square meter (kg/m^2).
2. Healthy as defined by:

   1. the absence of clinically significant illness and surgery within 4 weeks prior to study drug administration.
   2. the absence of clinically significant history of neurological, endocrine, cardiovascular, respiratory, hematological, immunological, psychiatric, gastrointestinal, renal, hepatic, and metabolic disease.
3. Female participants of non-childbearing potential must be:

   1. post-menopausal (spontaneous amenorrhea for at least 12 months prior to dosing) with confirmation by documented follicle-stimulating hormone (FSH) levels >=40 milli-international units per milliliter (mIU/mL); or
   2. surgically sterile (bilateral oophorectomy, bilateral salpingectomy, hysterectomy, or bilateral tubal occlusion) at least 3 months prior to dosing.
4. Participants must be willing not to donate sperm for 90 days or ova (egg) for 6 months after the last dose.
5. Sexually active females of childbearing potential and non-sterile males must be willing to use an acceptable contraceptive method throughout the study.
6. Able to understand the study procedures and provide signed informed consent to participate in the study.

Exclusion Criteria:

1. Any clinically significant abnormal finding at physical examination.
2. Clinically significant abnormal laboratory test results including biochemistry, hematology, urinalysis, and coagulation results, or positive serology test results for hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibody, or human immunodeficiency virus (HIV) antigen and antibody, or QuantiFERON®-TB test at screening.
3. Positive pregnancy test or lactating female participant.
4. Positive urine drug screen, urine cotinine test, or alcohol breath test at screening or Day -1.
5. History of significant allergic reactions (example, anaphylactic reaction, hypersensitivity, angioedema) to any drug.
6. Clinically significant ECG abnormalities or vital signs abnormalities (systolic blood pressure lower than 90 or over 140 millimetres of mercury (mmHg), diastolic blood pressure lower than 40 or over 90 mmHg, heart rate less than 40 or over 100 beats per minute (bpm), respiratory rate less than 10 or over 22 bpm), or oxygen saturation less than 95 percent (%) oxygen at screening.
7. History of drug abuse within 1 year prior to screening as determined by the investigator.
8. History of alcohol abuse within 1 year prior to screening or regular use of alcohol within 1 month prior to screening that exceeds 10 units of alcohol per week for women and men (1 unit = 375 [milliliter] mL of beer 3.5%, 100 mL of wine 13.5%, or 30 mL of distilled alcohol 40%).
9. History of active tuberculosis or presence of active or latent tuberculosis. Previous latent tuberculosis that has been treated and is no longer active is not exclusionary.
10. History of clinically significant opportunistic infection (example, invasive candidiasis or pneumocystis pneumonia).
11. History of serious local infection (example, cellulitis, abscess) or systemic infection (example, septicemia) within 3 months prior to screening.
12. Presence of fever (body temperature greater than (>) 37.5 degrees Celsius (°C) (example, a fever associated with a symptomatic viral or bacterial infection) within 2 weeks prior to dosing.
13. Use of medications within the timeframes specified.
14. Participation in a clinical research study involving the administration of an investigational or marketed drug or device within 30 days prior to the first dosing, administration of a biological product in the context of a clinical research study within 90 days prior to the first dosing, or simultaneous participation in an investigational study involving no drug or device administration.
15. Donation of plasma within 7 days prior to dosing or donation or loss of 500 mL or more of whole blood within 8 weeks prior to dosing.
16. Any reason which, in the opinion of the Investigator, would prevent the participant from participating in the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Estimated)
Dates: Start 2024-09-17 (Actual); Primary Completion 2025-02-27 (Estimated); Study Completion 2025-02-27 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events (AEs) | Up to final follow-up (SAD Part: up to 8 days: MAD Part: up to 14 days)
  An AE is defined as any untoward medical occurrence in a participant or clinical trial participant administered a pharmaceutical product and which does not necessarily have a causal relationship with the treatment. An AE can, therefore, be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not considered related to the medicinal (investigational) product. Any clinically significant changes in vital signs, electrocardiogram (ECG) measurement, physical examination and clinical laboratory parameters will be recorded as AE.

SECONDARY OUTCOMES:
SAD Part: Area under the concentration-time curve from time zero until the last observed concentration (AUC0-t) of H021 | pre-dose and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, and 48 hours post-dose
  AUC0-t is an area under the concentration-time curve from time zero (pre-dose) to time of last observed concentration.
SAD Part: Area under the concentration-time curve from time zero to infinity (AUC0-infinity) of H021 | pre-dose and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, and 48 hours post-dose
  AUC0-infinity is an area under the concentration-time curve from time zero to infinity (extrapolated).
SAD Part: Maximal observed concentration (Cmax) of H021 | pre-dose and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, and 48 hours post-dose
  Cmax is a measure of the maximum amount of drug in the plasma after the dose was given.
SAD Part: Time to Reach Cmax (Tmax) of H021 | pre-dose and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, and 48 hours post-dose
  Tmax is a measure of the time to reach the maximum concentration in the plasma after the dose was given.
SAD Part: Lag Time (Tlag) of H021 | pre-dose and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, and 48 hours post-dose
  Tlag is time of observation prior to the first observation with a measurable (non-zero) concentration (for food effect cohort only).
SAD Part: Residual area of H021 | pre-dose and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24), and 48 hours post-dose
  Residual area is calculated as percentage of AUC0-inf due to extrapolation from the time of the last observed concentration to infinity, calculated as [1 - (AUC0-t/AUC0-inf)] x 100.
SAD Part: Terminal elimination half-life (T1/2 el) of H021 | pre-dose and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, and 48 hours post-dose
  T1/2 el is defined as the duration until observation of half of the maximum concentration of drug dose.
SAD Part: Terminal elimination rate constant (Kel) of H021 | pre-dose and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, and 48 hours post-dose
  Kel is defined as first-order rate constant associated with the terminal (log-linear) portion of the curve.
SAD Part: Apparent clearance (CL/F) of H021 | pre-dose and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, and 48 hours post-dose
  CL/F is apparent total clearance of the drug from plasma after oral administration
SAD Part: Apparent volume of distribution (Vz/F) of H021 | pre-dose and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, and 48 hours post-dose
  Vz/F is apparent volume of distribution during terminal phase after non-intravenous administration
SAD Part: Cumulative Urinary Excretion From Time Zero to Time t (Ae0-t) of H021 | pre-dose (spot; within 2 hours) and 0-4, 4-8, 8-12, 12-24, and 24-48 hours post-dose
  Ae0-t is defined as cumulative urinary excretion from time zero to time t, calculated as the sum of the amounts excreted over each collection interval.
SAD Part: Maximal Rate of Urinary Excretion (Rmax) of H021 | pre-dose (spot; within 2 hours) and 0-4, 4-8, 8-12, 12-24, and 24-48 hours post-dose
  Rmax is defined as maximal rate of urinary excretion, calculated by dividing the amount of drug excreted in each collection interval by the time over which it was collected.
SAD Part: Time of Maximal Urinary Excretion (TRmax) of H021 | pre-dose (spot; within 2 hours) and 0-4, 4-8, 8-12, 12-24, and 24-48 hours post-dose
  TRmax is defined as time of maximal urinary excretion, calculated as the midpoint of the collection interval during which Rmax occurred.
SAD Part: Renal Clearance (CLR) of H021 | pre-dose (spot; within 2 hours) and 0-4, 4-8, 8-12, 12-24, and 24-48 hours post-dose
  CLR is renal clearance, calculated as Ae0-t /AUC0-t.
MAD Part: Area under the concentration-time curve from time zero to time 24 hours (AUC0-24) of H021 | Day 1 at pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48 hours post-first dose; predose on Days 4, 5, 6; Day 7 at predose and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48 hours post-last dose
  AUC0-24 is an area under the concentration-time curve from time zero to 24 hours post-dose.
MAD Part: Cmax of H021 | Day 1 at pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48 hours post-first dose; predose on Days 4, 5, 6; Day 7 at predose and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48 hours post-last dose
  Cmax is a measure of the maximum amount of drug in the plasma after the dose was given.
MAD Part: Tmax of H021 | Day 1 at pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48 hours post-first dose; predose on Days 4, 5, 6; Day 7 at predose and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48 hours post-last dose
  Tmax is a measure of the time to reach the maximum concentration in the plasma after the dose was given.
MAD Part: Area under the concentration-time curve for one dosing interval (τ) at steady- state (AUC0-τ) of H021 | Day 1 at pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48 hours post-first dose; predose on Days 4, 5, 6; Day 7 at predose and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48 hours post-last dose
  AUC0-τ is an area under the concentration-time curve for one dosing interval (τ) at steady- state. In this study τ = 24 hours (equivalent to AUC0-24) will be reported.
MAD Part: Cmax ss of H021 | Day 1 at pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48 hours post-first dose; predose on Days 4, 5, 6; Day 7 at predose and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48 hours post-last dose
  Cmax ss is a measure of the maximum amount of drug in the plasma at steady-state after the dose was given.
MAD Part: Tmax ss of H021 | Day 1 at pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48 hours post-first dose; predose on Days 4, 5, 6; Day 7 at predose and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48 hours post-last dose
  Tmax ss is a measure of the time to reach the maximum concentration in the plasma at steady state after the dose was given.
MAD Part: Minimal observed concentration at steady-state (Cmin ss) of H021 | Day 1 at pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48 hours post-first dose; predose on Days 4, 5, 6; Day 7 at predose and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48 hours post-last dose
  Cmin ss is minimal observed concentration at steady-state.
MAD Part: AUC0-t of H021 | Day 1 at pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48 hours post-first dose; predose on Days 4, 5, 6; Day 7 at predose and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48 hours post-last dose
  AUC0-t is an area under the concentration-time curve from time zero (pre-dose) to time of last observed concentration.
MAD Part: AUC0-inf of H021 | Day 1 at pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48 hours post-first dose; predose on Days 4, 5, 6; Day 7 at predose and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48 hours post-last dose
  AUC0-infinity is an area under the concentration-time curve from time zero to infinity (extrapolated).
MAD Part: Residual area of H021 | Day 1 at pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48 hours post-first dose; predose on Days 4, 5, 6; Day 7 at predose and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48 hours post-last dose
  Residual area is calculated as percentage of AUC0-inf due to extrapolation from the time of the last observed concentration to infinity, calculated as [1 - (AUC0-t/AUC0-inf)] x 100.
MAD Part: T½ el of H021 | Day 1 at pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48 hours post-first dose; predose on Days 4, 5, 6; Day 7 at predose and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48 hours post-last dose
  T1/2 el is defined as the duration until observation of half of the maximum concentration of drug dose.
MAD Part: Kel of H021 | Day 1 at pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48 hours post-first dose; predose on Days 4, 5, 6; Day 7 at predose and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48 hours post-last dose
  Kel is defined as first-order rate constant associated with the terminal (log-linear) portion of the curve.
MAD Part: Apparent clearance at steady-state (Clss/F) of H021 | Day 1 at pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48 hours post-first dose; predose on Days 4, 5, 6; Day 7 at predose and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48 hours post-last dose
  Clss/F is apparent clearance at steady-state.
MAD Part: Apparent volume of distribution at steady-state (Vz ss/F) of H021 | Day 1 at pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48 hours post-first dose; predose on Days 4, 5, 6; Day 7 at predose and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48 hours post-last dose
  Vz ss/F is apparent volume of distribution at steady-state.
MAD Part: Accumulation ratio (RAUC) | Day 1 at pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48 hours post-first dose; predose on Days 4, 5, 6; Day 7 at predose and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48 hours post-last dose
  RAUC is accumulation ratio for AUC.
MAD Part: Accumulation Ratio (RCmax) | Day 1 at pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48 hours post-first dose; predose on Days 4, 5, 6; Day 7 at pre-dose and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48 hours post-last dose
  RCmax is accumulation ratio for Cmax.

OTHER OUTCOMES:
MAD Part: Change From Baseline in Micro-RNA-124 (miR-124) Expression in Peripheral Blood Mononuclear Cells (PBMCs) | Day 1 at predose, and at 12 hours, on Day 5 at predose, and on Day 7 at predose, and at 12 hours post-last dose
  Change from baseline in miR-124 expression in PBMCs will be assessed.
MAD Part: Change From Baseline in Interleukin (IL)-6, Tumor Necrosis Factor Alpha (TNF-α), IL-17A, and Interferon Gamma (IFN-γ) in Blood Serum | Day 1 at predose, and at 12 hours, on Day 5 at predose, and on Day 7 at predose, and at 12 hours post-last dose
  Change from baseline in IL-6, TNF-α, IL-17A, and IFN-γ in blood serum will be assessed.

CONTACTS AND LOCATIONS:
Locations (1):
- Nucleus Network Ply Ltd., Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No